CLINICAL TRIAL: NCT06900959
Title: Transcranial Static Field Stimulation (tSMS) and Transcranial Direct Current Stimulation (tDCS) for the Treatment of Neurological Symptoms
Acronym: NIBS-tSMS/tDCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Diego Centonze, MD, PhD, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIBS-tSMS/tDCS
Record Dates: First submitted 2025-03-11; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Neurological Diseases or Conditions
Keywords: neuromodulation; non-invasive brain stimulation; transcranial direct current stimulation tDCS; transcranial static field stimulation tSMS
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tSMS real and tDCS real (Experimental): * Real transcranial static magnetic field stimulation (tSMS): will be used to perform the experimental intervention in combination with transcranial Direct Current Stimulation (tDCS), with no interruption between the tSMS and tDCS. Expert personnel will administer 30-minute tSMS stimulations immediately before the tDCS stimulation. tSMS is a non-invasive brain stimulation (NIBS) technique that involves the application of a neodymium magnet to the scalp. Since the first study introducing this method, several others have confirmed that tSMS can lead to a reduction in corticospinal excitability.
  * Real transcranial Direct Current Stimulation (tDCS): This device will be used to perform the experimental intervention in combination with tSMS. tDCS stimulations, lasting 20 minutes, will be administered immediately following the tSMS stimulation. tDCS involves the application of weak electrical currents capable of generating an electric field that can modulate neural activity.
  Interventions: Combination Product: transcranial static field stimulation (tSMS) and transcranial (tDCS)
- tSMS real and tDCS sham (Active Comparator): * Real transcranial static magnetic field stimulation (tSMS): will be used to perform the experimental intervention in combination with transcranial Direct Current Stimulation (tDCS), with no interruption between the tSMS and tDCS. Expert personnel will administer 30-minute tSMS stimulations immediately before the tDCS stimulation. tSMS is a non-invasive brain stimulation (NIBS) technique that involves the application of a neodymium magnet to the scalp. Since the first study introducing this method, several others have confirmed that tSMS can lead to a reduction in corticospinal excitability.
  * Sham transcranial Direct Current Stimulation (tDCS): in the sham tDCS groups, the duration and electrodes application were the same to real tDCS, but the current was stopped 30 s thereafter. The subject felt the initial itching sensation, but no changes in cortical excitability are producedcapable of generating an electric field that can modulate neural activity.
  Interventions: Combination Product: transcranial static field stimulation (tSMS) and transcranial (tDCS)
- tSMS sham tDCS real (Active Comparator): * Sham transcranial static magnetic field stimulation (tSMS): in the sham tSMS groups, the duration and application of the device were the same as in the real tSMS, but the neodymium magnet is not placed at the location where it should be, and therefore, no actual stimulation occurs.
  * Real transcranial direct current stimulation (tDCS): will be administered immediately following the sham tSMS. tDCS stimulations, lasting 20 minutes, will be administered immediately following the tSMS stimulation. tDCS involves the application of weak electrical currents capable of generating an electric field that can modulate neural activity.
  Interventions: Combination Product: transcranial static field stimulation (tSMS) and transcranial (tDCS)
- tSMS sham tDCS sham (Sham Comparator): * Sham transcranial static magnetic field stimulation (tSMS): in the sham tSMS groups, the duration and application of the device were the same as in the real tSMS, but the neodymium magnet is not placed at the location where it should be, and therefore, no actual stimulation occurs.
  * Sham transcranial Direct Current Stimulation (tDCS): in the sham tDCS groups, the duration and electrodes application were the same to real tDCS, but the current was stopped 30 s thereafter. The subject felt the initial itching sensation, but no changes in cortical excitability are producedcapable of generating an electric field that can modulate neural activity.
  Interventions: Combination Product: transcranial static field stimulation (tSMS) and transcranial (tDCS)

INTERVENTIONS:
Combination Product: transcranial static field stimulation (tSMS) and transcranial (tDCS) — * tSMS is a non-invasive brain stimulation (NIBS) technique that involves the application of a neodymium magnet to the scalp. Since the initial study introducing this method, numerous subsequent studies have confirmed that tSMS can lead to a reduction in corticospinal excitability.
  * Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation (NIBS) technique that applies low-voltage electrical currents through surface electrodes on the scalp. Depending on the stimulation type (anodal or cathodal) tDCS can induce long-lasting increases or decreases in neuronal excitability and vascular-neuronal activity coupling. Cathodal stimulation leads to hyperpolarization and a reduction in excitability, whereas anodal stimulation induces depolarization and enhances excitability.

SUMMARY:
The presence of damage to the central and/or peripheral nervous system resulting from various pathologies, such as Multiple Sclerosis (MS), Amyotrophic Lateral Sclerosis (ALS), Parkinson's disease (PD), Alzheimer's disease (AD), dementia, traumatic brain injury (TBI), stroke, or other neurological syndromes, is commonly a cause of both physical and mental disability. This leads to symptoms in the patient, including: pain, migraines, headaches, neuropathic pain, trigeminal neuralgia, depression, anxiety, apathy, fatigue, cognitive decline, aphasia, functional motor disorders (FMD), neuromuscular tone alterations, and hyposthenia, in addition to involvement of various cognitive functions, such as decision-making, problem-solving, learning, memory, executive functions, social cognition, and emotional cognition. The presence of these neurological symptoms is often evident in a first clinical examination and is one of the main reasons for further healthcare consultations. These difficulties have a profound impact on the quality of life, affecting work, social, and family functioning.

In recent years, several non-invasive brain stimulation (NIBS) techniques have emerged, aimed at eliciting brain neural networks, such as transcranial static magnetic field stimulation (tSMS) and transcranial direct current stimulation (tDCS).

tSMS is an NIBS technique that involves the application of a neodymium magnet on the scalp. Since the first study proposing this method, several others have confirmed that tSMS can reduce corticospinal excitability. tDCS involves the application of weak electrical currents capable of generating an electric field that can modulate neural activity in an excitatory or inhibitory manner. NIBS techniques can be used experimentally to modulate cortical activity.

The primary aim of this proposal is to address the impact of neurological symptoms through the combination of tSMS with tDCS and rehabilitation techniques. Specifically, it aims to understand whether the combination of these neuromodulatory therapeutic NIBS methods can enhance symptom improvement in patients with neurological conditions.

To assess the impact of this intervention, a series of tests and questionnaires, described in detail below, will be used to evaluate the severity of the reported symptoms and secondary outcomes.

Moreover, the contribution of specific brain areas to the symptom will be evaluated through the direct modulation of brain activity. This modulation will be achieved using an additional NIBS technique, such as Transcranial Magnetic Stimulation (TMS). TMS, in particular, is a non-invasive method for stimulating neurons in the brain's superficial areas, which has been frequently used in neurology as a diagnostic and research tool since its introduction. TMS uses magnetic fields to induce electrical currents capable of facilitating or inhibiting cortical activity.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged between 18 and 80 years;
* Presence of a neurological disorder, specifically the following conditions will be considered: MS, ALS, PD, AD, Dementias, TBI, neurosurgical interventions, stroke, fibromyalgia, epilepsy, headache, migraine, with at least one of the following symptoms: pain, neuropathic pain, neuralgias, depression, anxiety, apathy, fatigue, cognitive decline, aphasia, functional motor disorders (FMD), neuromuscular tone alterations, hyposthenia, involvement of multiple cognitive functions (including decision-making, problem-solving, learning, memory, executive functions, social and emotional cognition);
* Patients must be able to follow the protocol instructions for the duration of the study;
* Be able to understand the purposes and risks of the study;
* Be able to understand and provide written informed consent to the study.

Exclusion Criteria:

* Partial or total inability to understand or make decisions, inability to provide written informed consent for the study;
* Patients with a history or presence of any unstable medical condition, such as neoplasms or infections;
* Women with a positive pregnancy test at baseline or planning to become pregnant. Women who are breastfeeding or have given birth within the last three months prior to the start of the study;
* Use of medications that increase the risk of seizures (e.g., Fampridine, 4-aminopyridine);
* Concurrent use of medications that may alter synaptic transmission and plasticity (L-dopa, antiepileptics);
* In the case of using NIBS techniques, subjects should not have any contraindications specific to this method (for further details, see the "Methods" and the "Stimulation Assessment Questionnaire" attached to this proposal).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-11 (Estimated); Primary Completion 2025-12-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline at one week
  The VAS is a self-administered scale in which patients indicate the intensity of pain experienced by selecting a point on a continuous line ranging from 0 to 100 mm, representing the absence of pain to the worst pain, respectively.

SECONDARY OUTCOMES:
Neurological clinical assessment through the Expanded Disability Status Scale (EDSS) | Change from baseline at one month
  The Expanded Disability Status Scale (EDSS) is a clinician-administered assessment scale evaluating the functional systems of the central nervous system. The EDSS is used to describe disease progression in patients with multiple sclerosis MS and to assess the effectiveness of therapeutic interventions in clinical trials. It consists of ordinal rating system ranging from 0 (normal neurological status) to 10 (death due to MS) in 0.5 increments interval (when reaching EDSS 1).
Measurement of motor cortex plasticity through transcranial magnetic stimulation (TMS) | Change from baseline at one month
  Measurement of motor cortex plasticity (iTBS) through transcranial magnetic stimulation (TMS). The mean amplitudes of motor evoked potentials (MEP) will be recorded following iTBS, at each time point after iTBS (5, 15, and 30 minutes). The LTP-like effect will be expressed as percentage changes relative to the baseline MEPs.
Explore the effects of tSMS+tDCS treatment through the collection of biological material (blood and plasma) | Change from baseline at one month
  The blood samples, immediately after collection, will undergo the necessary procedures for isolating the different components. These will then be used to analyze the levels of microRNA, cytokines, chemokines, cellular growth factors, markers of neuronal damage (tau, phosphorylated and truncated tau, neurofilaments), mitochondrial markers (lactate), and free d-amino acids. Genotyping studies will be conducted to identify single nucleotide polymorphisms (SNPs) in coding and/or regulatory regions of genes (microRNA or protein) that correlate with specific clinical parameters and the levels of the identified potential biomarkers.
Brief Pain Inventory (BPI) | Change from baseline at one month
  The Brief Pain Inventory (BPI) is a self-administered measure of the sensory and reactive dimensions of pain that is the severity or intensity of the pain and the level of interference it has on various aspects of life. Interference is divided into activity and affective sub-dimensions. The BPI starts with a screening question, asking about the presence of pain and a body chart is used to indicate painful regions as well as the worst region. These items have not been evaluated. This is followed by the core BPI items: the rating scales for pain severity and interference. Numerical rating scales from 0 to 10 are used for all items. The anchors for pain severity scales are 0 = 'no pain' and 10 = 'pain as bad as you can imagine', whilst the interference anchors are 0 = 'no interference' and 10 = 'interferes completely'.
Zung Self-Rating Anxiety Scale (SAS) | Change from baseline at one month
  The Zung Self-Rating Anxiety Scale (SAS) is a 20-item self-report assessment device built to measure anxiety levels.
  The total raw scores range from 20 to 80:
  * 20-44 Normal Range
  * 45-59 Mild to Moderate Anxiety Levels
  * 60-74 Marked to Severe Anxiety Levels
  * 75 and above Extreme Anxiety Levels
Zung Self-Rating Depression Scale (SDS) | Change from baseline at one month
  The Zung Self-Rating Depression Scale (SDS) is a short self-administered survey to quantify the depressed status of a patient. There are 20 items on the scale that rate the four common characteristics of depression: the pervasive effect, the physiological equivalents, other disturbances, and psychomotor activities. There are ten positively worded and ten negatively worded questions. Each question is scored on a scale of 1-4 (a little of the time, some of the time, good part of the time, most of the time).
  The scores range from 25-100.
  * 25-49 Normal Range
  * 50-59 Mildly Depressed
  * 60-69 Moderately Depressed
  * 70 and above Severely Depressed
The Pittsburgh Sleep Quality Index (PSQI) | Change from baseline at one month
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
The Short Form 36 Health Survey (SF-36) | Change from baseline at one month
  The Short Form (36) Health Survey (SF-36) is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability, a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
The Beck Depression Inventory (BDI-II) | Change from baseline at one month
  The Beck Depression Inventory (BDI-II) is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs are the following:
  * 0-13: minimal depression
  * 14-19: mild depression
  * 20-28: moderate depression
  * 29-63: severe depression.
State-Trait Anxiety Inventory (STAI) | Change from baseline at one month
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Each type of anxiety has its own scale of 20 different questions that are scored. Scores range from 20 to 80, higher scores are positively correlated with higher levels of anxiety.
The Toronto Alexithymia Scale (TAS-20) | Change from baseline at one month
  The Toronto Alexithymia Scale (TAS-20) is a measure of deficiency in understanding, processing, or describing emotions. The current version has twenty statements rated on a five-point Likert scale. The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale.
The Fibromyalgia Impact Questionnaire (FIQ) | Change from baseline at one month
  The Fibromyalgia Impact Questionnaire (FIQ) is a brief 10-item, self-administered instrument that measures physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well being. The FIQ is composed of 10 items. The first item contains 11 questions related to physical functioning - each question is rated on a 4 point Likert type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. Items 4 through 10 are horizontal linear scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety and depression. The FIQ is composed of ten questions with a maximum score of 100, higher scores reflecting greater impact.
Modified Fatigue Impact Scale (MFIS) | Change from baseline at one month
  The Modified Fatigue Impact Scale (MFIS) provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning.Items on the MFIS can be aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities.
  * Physical Subscale: this scale can range from 0 to 36. It is computed by adding raw scores on the following items: 4+6+7+10+13+14+17+20+21.
  * Cognitive Subscale: this scale can range from 0 to 40. It is computed by adding raw scores on the following items: 1+2+3+5+11+12+15+16+18+19.
  * Psychosocial Subscale: this scale can range from 0 to 8. It is computed by adding raw scores on the following items: 8+9.
  * Total MFIS Score: the total MFIS score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales
The Multiple Sclerosis Impact Scale (MSIS-29) | Change from baseline at one month
  The Multiple Sclerosis Impact Scale (MSIS-29) is a 29-item self-report measure comprised of 20 items associated with a physical scale and 9 items associated with a psychological scale.1 Items question patients (or their proxies) about the impact of multiple sclerosis (MS) on day-to-day life in the last 2 weeks. All items have 5 response options from 1 (not at all) to 5 (extremely). Each of the 2 scales are scored by summing the responses across items, then converting to a 0 to 100 scale, where 100 indicates greater impact of disease on daily function (worse health).
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Change from baseline at one month
  The Multiple Sclerosis Quality of Life-54 (MSQOL-54) is a multidimensional health-related quality of life measure that combines both generic and multiple sclerosis MS-specific items into a single instrument. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The summary scores are the physical health composite summary and the mental health composite summary. The single item measures are satisfaction with sexual function and change in health. The 54 items are divided into 12 multi-item and 2 single-item scales. The MSQOL-54 items are transformed linearly to 0-100 scores, and final scores are obtained by averaging items within the scales.
Fatigue severity scale (FSS) | Change from baseline at one month
  The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities. It is simple to understand and takes an average of eight minutes to answer

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Neurologico Mediterraneo IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zitser J, Allen IE, Falgas N, Le MM, Neylan TC, Kramer JH, Walsh CM. Pittsburgh Sleep Quality Index (PSQI) responses are modulated by total sleep time and wake after sleep onset in healthy older adults. PLoS One. 2022 Jun 24;17(6):e0270095. doi: 10.1371/journal.pone.0270095. eCollection 2022. PMID 35749529
- [Result] Zhang R, Lam CLM, Peng X, Zhang D, Zhang C, Huang R, Lee TMC. Efficacy and acceptability of transcranial direct current stimulation for treating depression: A meta-analysis of randomized controlled trials. Neurosci Biobehav Rev. 2021 Jul;126:481-490. doi: 10.1016/j.neubiorev.2021.03.026. Epub 2021 Mar 28. PMID 33789158
- [Result] Zettin M, Bondesan C, Nada G, Varini M, Dimitri D. Transcranial Direct-Current Stimulation and Behavioral Training, a Promising Tool for a Tailor-Made Post-stroke Aphasia Rehabilitation: A Review. Front Hum Neurosci. 2021 Dec 20;15:742136. doi: 10.3389/fnhum.2021.742136. eCollection 2021. PMID 34987366
- [Result] Wilson MA, Greenwell D, Meek AW, Poston B, Riley ZA. Neuroenhancement of a dexterous motor task with anodal tDCS. Brain Res. 2022 Sep 1;1790:147993. doi: 10.1016/j.brainres.2022.147993. Epub 2022 Jun 26. PMID 35760153
- [Result] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- [Result] Verhoog MB, Goriounova NA, Obermayer J, Stroeder J, Hjorth JJ, Testa-Silva G, Baayen JC, de Kock CP, Meredith RM, Mansvelder HD. Mechanisms underlying the rules for associative plasticity at adult human neocortical synapses. J Neurosci. 2013 Oct 23;33(43):17197-208. doi: 10.1523/JNEUROSCI.3158-13.2013. PMID 24155324
- [Result] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Result] Vanbellingen T, Nyffeler T, Nigg J, Janssens J, Hoppe J, Nef T, Muri RM, van Wegen EEH, Kwakkel G, Bohlhalter S. Home based training for dexterity in Parkinson's disease: A randomized controlled trial. Parkinsonism Relat Disord. 2017 Aug;41:92-98. doi: 10.1016/j.parkreldis.2017.05.021. Epub 2017 May 25. PMID 28578819
- [Result] Taghizadeh G, Sarlak N, Fallah S, Sharabiani PTA, Cheraghifard M. Minimal clinically important differenceof fatigue severity scale in patients with chronic stroke. J Stroke Cerebrovasc Dis. 2024 Apr;33(4):107577. doi: 10.1016/j.jstrokecerebrovasdis.2024.107577. Epub 2024 Jan 12. PMID 38325034
- [Result] Strijbis EM, Repovic P, Mostert J, Bowen JD, Uitdehaag BM, Cutter G, Koch MW. The MSIS-29 and SF-36 as outcomes in secondary progressive MS trials. Mult Scler. 2022 Sep;28(10):1606-1619. doi: 10.1177/13524585221105465. PMID 35876467
- [Result] Soto-Leon V, Torres-Llacsa M, Mordillo-Mateos L, Carrasco-Lopez C, Pineda-Pardo JA, Velasco AI, Abad-Toribio L, Tornero J, Foffani G, Strange BA, Oliviero A. Static magnetic field stimulation over motor cortex modulates resting functional connectivity in humans. Sci Rep. 2022 May 12;12(1):7834. doi: 10.1038/s41598-022-11859-5. PMID 35551490
- [Result] Somaa FA, de Graaf TA, Sack AT. Transcranial Magnetic Stimulation in the Treatment of Neurological Diseases. Front Neurol. 2022 May 20;13:793253. doi: 10.3389/fneur.2022.793253. eCollection 2022. PMID 35669870
- [Result] Smirni D, Oliveri M, Misuraca E, Catania A, Vernuccio L, Picciolo V, Inzerillo F, Barbagallo M, Cipolotti L, Turriziani P. Verbal Fluency in Mild Alzheimer's Disease: Transcranial Direct Current Stimulation over the Dorsolateral Prefrontal Cortex. J Alzheimers Dis. 2021;81(3):1273-1283. doi: 10.3233/JAD-210003. PMID 33935089
- [Result] Sagliano L, D'Olimpio F, Panico F, Gagliardi S, Trojano L. The role of the dorsolateral prefrontal cortex in early threat processing: a TMS study. Soc Cogn Affect Neurosci. 2016 Dec;11(12):1992-1998. doi: 10.1093/scan/nsw105. Epub 2016 Aug 10. PMID 27510494
- [Result] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Result] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Result] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Result] Rooney S, McFadyen DA, Wood DL, Moffat DF, Paul PL. Minimally important difference of the fatigue severity scale and modified fatigue impact scale in people with multiple sclerosis. Mult Scler Relat Disord. 2019 Oct;35:158-163. doi: 10.1016/j.msard.2019.07.028. Epub 2019 Jul 28. PMID 31400557
- [Result] Poquet N, Lin C. The Brief Pain Inventory (BPI). J Physiother. 2016 Jan;62(1):52. doi: 10.1016/j.jphys.2015.07.001. Epub 2015 Aug 21. No abstract available. PMID 26303366
- [Result] Pereira LS, Muller VT, da Mota Gomes M, Rotenberg A, Fregni F. Safety of repetitive transcranial magnetic stimulation in patients with epilepsy: A systematic review. Epilepsy Behav. 2016 Apr;57(Pt A):167-176. doi: 10.1016/j.yebeh.2016.01.015. Epub 2016 Mar 10. PMID 26970993
- [Result] Pena-Gomez C, Sala-Lonch R, Junque C, Clemente IC, Vidal D, Bargallo N, Falcon C, Valls-Sole J, Pascual-Leone A, Bartres-Faz D. Modulation of large-scale brain networks by transcranial direct current stimulation evidenced by resting-state functional MRI. Brain Stimul. 2012 Jul;5(3):252-263. doi: 10.1016/j.brs.2011.08.006. Epub 2011 Sep 5. PMID 21962981
- [Result] Oliviero A, Mordillo-Mateos L, Arias P, Panyavin I, Foffani G, Aguilar J. Transcranial static magnetic field stimulation of the human motor cortex. J Physiol. 2011 Oct 15;589(Pt 20):4949-58. doi: 10.1113/jphysiol.2011.211953. Epub 2011 Aug 1. PMID 21807616
- [Result] Ochi M, Saeki S, Oda T, Matsushima Y, Hachisuka K. Effects of anodal and cathodal transcranial direct current stimulation combined with robotic therapy on severely affected arms in chronic stroke patients. J Rehabil Med. 2013 Feb;45(2):137-40. doi: 10.2340/16501977-1099. PMID 23306448
- [Result] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Result] Nitsche MA, Paulus W. Transcranial direct current stimulation--update 2011. Restor Neurol Neurosci. 2011;29(6):463-92. doi: 10.3233/RNN-2011-0618. PMID 22085959
- [Result] Nielsen G, Stone J, Matthews A, Brown M, Sparkes C, Farmer R, Masterton L, Duncan L, Winters A, Daniell L, Lumsden C, Carson A, David AS, Edwards M. Physiotherapy for functional motor disorders: a consensus recommendation. J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1113-9. doi: 10.1136/jnnp-2014-309255. Epub 2014 Nov 28. PMID 25433033
- [Result] Naegel S, Biermann J, Theysohn N, Kleinschnitz C, Diener HC, Katsarava Z, Obermann M, Holle D. Polarity-specific modulation of pain processing by transcranial direct current stimulation - a blinded longitudinal fMRI study. J Headache Pain. 2018 Oct 24;19(1):99. doi: 10.1186/s10194-018-0924-5. PMID 30355321
- [Result] Mori F, Rossi S, Piccinin S, Motta C, Mango D, Kusayanagi H, Bergami A, Studer V, Nicoletti CG, Buttari F, Barbieri F, Mercuri NB, Martino G, Furlan R, Nistico R, Centonze D. Synaptic plasticity and PDGF signaling defects underlie clinical progression in multiple sclerosis. J Neurosci. 2013 Dec 4;33(49):19112-9. doi: 10.1523/JNEUROSCI.2536-13.2013. PMID 24305808
- [Result] Matsumoto T, Watanabe T, Ito K, Horinouchi T, Shibata S, Kurumadani H, Sunagawa T, Mima T, Kirimoto H. Effect of transcranial static magnetic stimulation over unilateral or bilateral motor association cortex on performance of simple and choice reaction time tasks. Front Hum Neurosci. 2023 Dec 4;17:1298761. doi: 10.3389/fnhum.2023.1298761. eCollection 2023. PMID 38111674
- [Result] Marangolo P, Fiori V, Campana S, Calpagnano MA, Razzano C, Caltagirone C, Marini A. Something to talk about: enhancement of linguistic cohesion through tdCS in chronic non fluent aphasia. Neuropsychologia. 2014 Jan;53:246-56. doi: 10.1016/j.neuropsychologia.2013.12.003. Epub 2013 Dec 11. PMID 24333381
- [Result] Luo Y, Yang W, Li N, Yang X, Zhu B, Wang C, Hou W, Wang X, Wen H, Tian X. Anodal Transcranial Direct Current Stimulation Can Improve Spatial Learning and Memory and Attenuate Abeta42 Burden at the Early Stage of Alzheimer's Disease in APP/PS1 Transgenic Mice. Front Aging Neurosci. 2020 May 13;12:134. doi: 10.3389/fnagi.2020.00134. eCollection 2020. PMID 32595486
- [Result] Longo V, Barbati SA, Re A, Paciello F, Bolla M, Rinaudo M, Miraglia F, Alu F, Di Donna MG, Vecchio F, Rossini PM, Podda MV, Grassi C. Transcranial Direct Current Stimulation Enhances Neuroplasticity and Accelerates Motor Recovery in a Stroke Mouse Model. Stroke. 2022 May;53(5):1746-1758. doi: 10.1161/STROKEAHA.121.034200. Epub 2022 Mar 16. PMID 35291824
- [Result] Liu CS, Rau A, Gallagher D, Rajji TK, Lanctot KL, Herrmann N. Using transcranial direct current stimulation to treat symptoms in mild cognitive impairment and Alzheimer's disease. Neurodegener Dis Manag. 2017 Oct;7(5):317-329. doi: 10.2217/nmt-2017-0021. Epub 2017 Oct 18. PMID 29043928
- [Result] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230
- [Result] Li S, Zhang B, Guo Y, Zhang J. The association between alexithymia as assessed by the 20-item Toronto Alexithymia Scale and depression: A meta-analysis. Psychiatry Res. 2015 May 30;227(1):1-9. doi: 10.1016/j.psychres.2015.02.006. Epub 2015 Feb 19. PMID 25769520
- [Result] Leite Silva ABR, Goncalves de Oliveira RW, Diogenes GP, de Castro Aguiar MF, Sallem CC, Lima MPP, de Albuquerque Filho LB, Peixoto de Medeiros SD, Penido de Mendonca LL, de Santiago Filho PC, Nones DP, da Silva Cardoso PMM, Ribas MZ, Galvao SL, Gomes GF, Bezerra de Menezes AR, Dos Santos NL, Mororo VM, Duarte FS, Dos Santos JCC. Premotor, nonmotor and motor symptoms of Parkinson's Disease: A new clinical state of the art. Ageing Res Rev. 2023 Feb;84:101834. doi: 10.1016/j.arr.2022.101834. Epub 2022 Dec 26. PMID 36581178
- [Result] Lee M. Clinimetrics: The Revised Fibromyalgia Impact Questionnaire. J Physiother. 2021 Jul;67(3):220-221. doi: 10.1016/j.jphys.2020.09.002. Epub 2020 Sep 25. No abstract available. PMID 32988791
- [Result] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Result] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818
- [Result] Knowles KA, Olatunji BO. Specificity of trait anxiety in anxiety and depression: Meta-analysis of the State-Trait Anxiety Inventory. Clin Psychol Rev. 2020 Dec;82:101928. doi: 10.1016/j.cpr.2020.101928. Epub 2020 Oct 10. PMID 33091745
- [Result] Knotkova H, Hamani C, Sivanesan E, Le Beuffe MFE, Moon JY, Cohen SP, Huntoon MA. Neuromodulation for chronic pain. Lancet. 2021 May 29;397(10289):2111-2124. doi: 10.1016/S0140-6736(21)00794-7. PMID 34062145
- [Result] Ilic TV, Meintzschel F, Cleff U, Ruge D, Kessler KR, Ziemann U. Short-interval paired-pulse inhibition and facilitation of human motor cortex: the dimension of stimulus intensity. J Physiol. 2002 Nov 15;545(1):153-67. doi: 10.1113/jphysiol.2002.030122. PMID 12433957
- [Result] Hsu WY, Cheng CH, Zanto TP, Gazzaley A, Bove RM. Effects of Transcranial Direct Current Stimulation on Cognition, Mood, Pain, and Fatigue in Multiple Sclerosis: A Systematic Review and Meta-Analysis. Front Neurol. 2021 Mar 8;12:626113. doi: 10.3389/fneur.2021.626113. eCollection 2021. PMID 33763014
- [Result] Huang YZ, Lu MK, Antal A, Classen J, Nitsche M, Ziemann U, Ridding M, Hamada M, Ugawa Y, Jaberzadeh S, Suppa A, Paulus W, Rothwell J. Plasticity induced by non-invasive transcranial brain stimulation: A position paper. Clin Neurophysiol. 2017 Nov;128(11):2318-2329. doi: 10.1016/j.clinph.2017.09.007. Epub 2017 Sep 28. PMID 29040922
- [Result] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Result] Hou WH, Wang TY, Kang JH. The effects of add-on non-invasive brain stimulation in fibromyalgia: a meta-analysis and meta-regression of randomized controlled trials. Rheumatology (Oxford). 2016 Aug;55(8):1507-17. doi: 10.1093/rheumatology/kew205. Epub 2016 May 5. PMID 27150193
- [Result] Hiew S, Nguemeni C, Zeller D. Efficacy of transcranial direct current stimulation in people with multiple sclerosis: a review. Eur J Neurol. 2022 Feb;29(2):648-664. doi: 10.1111/ene.15163. Epub 2021 Nov 19. PMID 34725881
- [Result] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Result] Heeren A, Billieux J, Philippot P, De Raedt R, Baeken C, de Timary P, Maurage P, Vanderhasselt MA. Impact of transcranial direct current stimulation on attentional bias for threat: a proof-of-concept study among individuals with social anxiety disorder. Soc Cogn Affect Neurosci. 2017 Feb 1;12(2):251-260. doi: 10.1093/scan/nsw119. PMID 27531388
- [Result] Hara Y. Brain plasticity and rehabilitation in stroke patients. J Nippon Med Sch. 2015;82(1):4-13. doi: 10.1272/jnms.82.4. PMID 25797869
- [Result] Guimaraes HC, Levy R, Teixeira AL, Beato RG, Caramelli P. Neurobiology of apathy in Alzheimer's disease. Arq Neuropsiquiatr. 2008 Jun;66(2B):436-43. doi: 10.1590/s0004-282x2008000300035. PMID 18641892
- [Result] van Groenestijn AC, Kruitwagen-van Reenen ET, Visser-Meily JM, van den Berg LH, Schroder CD. Associations between psychological factors and health-related quality of life and global quality of life in patients with ALS: a systematic review. Health Qual Life Outcomes. 2016 Jul 20;14(1):107. doi: 10.1186/s12955-016-0507-6. PMID 27439463
- [Result] Gonsalvez I, Spagnolo P, Dworetzky B, Baslet G. Neurostimulation for the treatment of functional neurological disorder: A systematic review. Epilepsy Behav Rep. 2021 Nov 9;16:100501. doi: 10.1016/j.ebr.2021.100501. eCollection 2021. PMID 34950864
- [Result] Giordano A, Testa S, Bassi M, Cilia S, Bertolotto A, Quartuccio ME, Pietrolongo E, Falautano M, Grobberio M, Niccolai C, Allegri B, Viterbo RG, Confalonieri P, Giovannetti AM, Cocco E, Grasso MG, Lugaresi A, Ferriani E, Nocentini U, Zaffaroni M, De Livera A, Jelinek G, Solari A, Rosato R. Assessing measurement invariance of MSQOL-54 across Italian and English versions. Qual Life Res. 2020 Mar;29(3):783-791. doi: 10.1007/s11136-019-02352-0. Epub 2019 Nov 9. PMID 31707695
- [Result] Giovagnoli AR, Paterlini C, Meneses RF, Martins da Silva A. Spirituality and quality of life in epilepsy and other chronic neurological disorders. Epilepsy Behav. 2019 Apr;93:94-101. doi: 10.1016/j.yebeh.2019.01.035. Epub 2019 Mar 6. PMID 30851485
- [Result] Gilmour GS, Nielsen G, Teodoro T, Yogarajah M, Coebergh JA, Dilley MD, Martino D, Edwards MJ. Management of functional neurological disorder. J Neurol. 2020 Jul;267(7):2164-2172. doi: 10.1007/s00415-020-09772-w. Epub 2020 Mar 19. PMID 32193596
- [Result] Ghahfarrokhi MM, Banitalebi E, Negaresh R, Motl RW. Home-Based Exercise Training in Multiple Sclerosis: A Systematic Review with Implications for Future Research. Mult Scler Relat Disord. 2021 Oct;55:103177. doi: 10.1016/j.msard.2021.103177. Epub 2021 Jul 27. PMID 34343867
- [Result] Garofalo S, di Pellegrino G. Individual differences in the influence of task-irrelevant Pavlovian cues on human behavior. Front Behav Neurosci. 2015 Jun 24;9:163. doi: 10.3389/fnbeh.2015.00163. eCollection 2015. PMID 26157371
- [Result] Forogh B, Rafiei M, Arbabi A, Motamed MR, Madani SP, Sajadi S. Repeated sessions of transcranial direct current stimulation evaluation on fatigue and daytime sleepiness in Parkinson's disease. Neurol Sci. 2017 Feb;38(2):249-254. doi: 10.1007/s10072-016-2748-x. Epub 2016 Oct 31. PMID 27796604
- [Result] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation for improving spasticity after stroke: A systematic review with meta-analysis. J Rehabil Med. 2016 Jul 18;48(7):565-70. doi: 10.2340/16501977-2097. PMID 27172484
- [Result] Ellis T, Motl RW. Physical activity behavior change in persons with neurologic disorders: overview and examples from Parkinson disease and multiple sclerosis. J Neurol Phys Ther. 2013 Jun;37(2):85-90. doi: 10.1097/NPT.0b013e31829157c0. PMID 23632452
- [Result] Dunstan DA, Scott N. Norms for Zung's Self-rating Anxiety Scale. BMC Psychiatry. 2020 Feb 28;20(1):90. doi: 10.1186/s12888-019-2427-6. PMID 32111187
- [Result] Dunstan DA, Scott N, Todd AK. Screening for anxiety and depression: reassessing the utility of the Zung scales. BMC Psychiatry. 2017 Sep 8;17(1):329. doi: 10.1186/s12888-017-1489-6. PMID 28886698
- [Result] Di Lazzaro V, Musumeci G, Boscarino M, De Liso A, Motolese F, Di Pino G, Capone F, Ranieri F. Transcranial static magnetic field stimulation can modify disease progression in amyotrophic lateral sclerosis. Brain Stimul. 2021 Jan-Feb;14(1):51-54. doi: 10.1016/j.brs.2020.11.003. Epub 2020 Nov 10. No abstract available. PMID 33186779
- [Result] De Vito F, Musella A, Fresegna D, Rizzo FR, Gentile A, Stampanoni Bassi M, Gilio L, Buttari F, Procaccini C, Colamatteo A, Bullitta S, Guadalupi L, Caioli S, Vanni V, Balletta S, Sanna K, Bruno A, Dolcetti E, Furlan R, Finardi A, Licursi V, Drulovic J, Pekmezovic T, Fusco C, Bruzzaniti S, Hornstein E, Uccelli A, Salvetti M, Matarese G, Centonze D, Mandolesi G. MiR-142-3p regulates synaptopathy-driven disease progression in multiple sclerosis. Neuropathol Appl Neurobiol. 2022 Feb;48(2):e12765. doi: 10.1111/nan.12765. Epub 2021 Oct 6. PMID 34490928
- [Result] De Icco R, Putorti A, De Paoli I, Ferrara E, Cremascoli R, Terzaghi M, Toscano G, Allena M, Martinelli D, Cosentino G, Grillo V, Colagiorgio P, Versino M, Manni R, Sances G, Sandrini G, Tassorelli C. Anodal transcranial direct current stimulation in chronic migraine and medication overuse headache: A pilot double-blind randomized sham-controlled trial. Clin Neurophysiol. 2021 Jan;132(1):126-136. doi: 10.1016/j.clinph.2020.10.014. Epub 2020 Nov 5. PMID 33271482
- [Result] Dayan E, Censor N, Buch ER, Sandrini M, Cohen LG. Noninvasive brain stimulation: from physiology to network dynamics and back. Nat Neurosci. 2013 Jul;16(7):838-44. doi: 10.1038/nn.3422. Epub 2013 Jun 25. PMID 23799477
- [Result] Davidson RJ, Irwin W. The functional neuroanatomy of emotion and affective style. Trends Cogn Sci. 1999 Jan;3(1):11-21. doi: 10.1016/s1364-6613(98)01265-0. PMID 10234222
- [Result] Cuerda-Ballester M, Martinez-Rubio D, Garcia-Pardo MP, Proano B, Cubero L, Calvo-Capilla A, Sancho-Cantus D, de la Rubia Orti JE. Relationship of Motor Impairment with Cognitive and Emotional Alterations in Patients with Multiple Sclerosis. Int J Environ Res Public Health. 2023 Jan 12;20(2):1387. doi: 10.3390/ijerph20021387. PMID 36674140
- [Result] Costanzo F, Menghini D, Maritato A, Castiglioni MC, Mereu A, Varuzza C, Zanna V, Vicari S. New Treatment Perspectives in Adolescents With Anorexia Nervosa: The Efficacy of Non-invasive Brain-Directed Treatment. Front Behav Neurosci. 2018 Jul 20;12:133. doi: 10.3389/fnbeh.2018.00133. eCollection 2018. PMID 30083095
- [Result] Campana S, Caltagirone C, Marangolo P. Combining Voxel-based Lesion-symptom Mapping (VLSM) With A-tDCS Language Treatment: Predicting Outcome of Recovery in Nonfluent Chronic Aphasia. Brain Stimul. 2015 Jul-Aug;8(4):769-76. doi: 10.1016/j.brs.2015.01.413. Epub 2015 Jan 30. PMID 25732786
- [Result] Cai M, Guo Z, Xing G, Peng H, Zhou L, Chen H, McClure MA, He L, Xiong L, He B, Du F, Mu Q. Transcranial Direct Current Stimulation Improves Cognitive Function in Mild to Moderate Alzheimer Disease: A Meta-Analysis. Alzheimer Dis Assoc Disord. 2019 Apr-Jun;33(2):170-178. doi: 10.1097/WAD.0000000000000304. PMID 31033517
- [Result] Brunoni AR, Moffa AH, Fregni F, Palm U, Padberg F, Blumberger DM, Daskalakis ZJ, Bennabi D, Haffen E, Alonzo A, Loo CK. Transcranial direct current stimulation for acute major depressive episodes: meta-analysis of individual patient data. Br J Psychiatry. 2016 Jun;208(6):522-31. doi: 10.1192/bjp.bp.115.164715. Epub 2016 Apr 7. PMID 27056623
- [Result] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Result] Brown L, Camarinos J. The Role of Physical Therapy in Concussion Rehabilitation. Semin Pediatr Neurol. 2019 Jul;30:68-78. doi: 10.1016/j.spen.2019.03.011. Epub 2019 Mar 27. PMID 31235023
- [Result] Beswick E, Forbes D, Johnson M, Newton J, Dakin R, Glasmcher S, Abrahams S, Carson A, Chandran S, Pal S. Non-motor symptoms in motor neuron disease: prevalence, assessment and impact. Brain Commun. 2023 Dec 7;6(1):fcad336. doi: 10.1093/braincomms/fcad336. eCollection 2024. PMID 38162906
- [Result] Bello-Haas VD. Physical therapy for individuals with amyotrophic lateral sclerosis: current insights. Degener Neurol Neuromuscul Dis. 2018 Jul 16;8:45-54. doi: 10.2147/DNND.S146949. eCollection 2018. PMID 30890895
- [Result] Begemann MJ, Brand BA, Curcic-Blake B, Aleman A, Sommer IE. Efficacy of non-invasive brain stimulation on cognitive functioning in brain disorders: a meta-analysis. Psychol Med. 2020 Nov;50(15):2465-2486. doi: 10.1017/S0033291720003670. Epub 2020 Oct 19. PMID 33070785
- [Result] Alashram AR, Annino G, Raju M, Padua E. Effects of physical therapy interventions on balance ability in people with traumatic brain injury: A systematic review. NeuroRehabilitation. 2020;46(4):455-466. doi: 10.3233/NRE-203047. PMID 32508337